CLINICAL TRIAL: NCT03702543
Title: Managing Vascular Dementia Risk Factors With SymTrend
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: SymTrend Inc. (Industry)
Collaborators: National Institute on Aging (NIA) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1R43AG060851-01 (NIH); 1R43AG060851-01 (NIH)
Record Dates: First submitted 2018-10-05; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Vascular Dementia
MeSH Terms: conditions — Dementia, Vascular

STUDY DESIGN:
Intervention Model Description: In this feasibility study, a customized electronic diary will be provided to collect data 1) from bluetooth devices, 2) from Apple Health app information, and 3) from self-reported diary information. Researchers will provide feedback via charts and reminders/text messages to encourage management of vascular risk factors.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: SymTrend, Inc. — Use of SymTrend and Apple Health apps with feedback and strategies provided.

SUMMARY:
Individuals with uncontrolled vascular disease are at risk for an insidious progression of brain injury starting in early to midlife and ultimately culminating in a vascular dementia, robbing them of activities of daily living independence. Successful containment of this progression requires rigorous vascular risk factor management - the control of blood pressure, blood sugars, weight, and alcohol consumption; the cessation of smoking, and an increase in aerobic activity. SymTrend's mobile and web system for managing vascular risk factors will help improve adherence to health and lifestyle strategies, will stem cognitive decline, and will preserve independence in the community for older adults.

DETAILED DESCRIPTION:
Neurologists from Massachusetts General Hospital will refer 10 adults with vascular mild cognitive impairment for participation in this project. The patients will be given Bluetooth devices appropriate for their condition and will be trained to use SymTrend and Apple Health software. They will use the software and devices for three months; will receive messages throughout from the system and/or a research coordinator about their progress, with encouragement and strategies to fully manage their symptoms; and their neurologist will be in communication with them about the progress charts and will adjust their care on the basis of this real-time data.

ELIGIBILITY:
Inclusion Criteria:

* Prior incidence of neurological event such as transient ischemic attack, stroke.

Exclusion Criteria:

* Inability to use smartphone,
* Inability to read English

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-10-14 (Estimated); Study Completion 2019-10-14 (Estimated)

PRIMARY OUTCOMES:
Improved management of blood sugar | three months
  Blood sugars are measured regularly and are maintained within bounds prescribed by MD
Improved blood pressure management | three months
  Blood pressure is measured regularly and is within bounds prescribed by MD
Reduced smoking | three months
  Number of cigarettes smoked is reduced or eliminated
Weight is reduced if necessary | three months
  Food intake is reduced and is healthier, and as a consequence weight is reduced
Activity level is increased | three months
  Step count increases continuously throughout study period

SECONDARY OUTCOMES:
Fatigue is reduced if originally is a problem | three months
  Hours sleep increases and frequency of sleep interruption reduces

CONTACTS AND LOCATIONS:
Overall Officials: Minna Levine, Phd, Principal Investigator — SymTrend Inc.
Locations (1):
- Neurology Department, Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No